CLINICAL TRIAL: NCT06046222
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study to Investigate the Efficacy and Safety of NS-229 in the Treatment of Eosinophilic Granulomatosis With Polyangiitis
Brief Title: Trial of Efficacy and Safety of NS-229 Versus Placebo in Patients With Eosinophilic Granulomatosis With Polyangiitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS229-P2-01
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-12

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis; Churg-Strauss Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NS-229 (Experimental): Self-administer NS-229 in consecutive 28 weeks.
  Interventions: Drug: NS-229
- Placebo (Placebo Comparator): Self-administer matching placebo in consecutive 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NS-229 — Experimental
  Arms: NS-229
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This study will enroll male and female subjects who are 18 years of age or older with Eosinophilic Granulomatosis With Polyangiitis.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind study is to investigate the efficacy and safety of NS229 compared with placebo over a 28-week study treatment period in subjects with Eosinophilic Granulomatosis with Polyangiitis (EGPA) receiving background corticosteroid therapy with or without Mepolizumab/Benralizumab therapy. During the treatment period corticosteroid dose will be tapered.

The key outcomes in the study focus on evaluation of clinical remission, defined as Birmingham Vasculitis Activity Score (BVAS)=0 with a corticosteroid dose of <=4 mg/day prednisolone/prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent prior to participation in the study.
* Male or female subjects aged ≥18 years at the time the informed consent form is signed.
* Diagnosis of EGPA: Subjects who have been diagnosed with EGPA based on the history or presence of eosinophilia plus at least a history or presence of 2 of additional features of EGPA.
* Subjects receive background OGC dose of ≥7.5 mg/day with or without stable treatment with Mepolizumab/Benralizumab.
* Use of adequate contraception.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Current diagnosis of either granulomatosis with polyangiitis or microscopic polyangiitis
* Imminently life-threatening EGPA at the time of screening.
* History or presence of any form of cancer within 5 years prior to screening.
* Serious liver, renal, blood, or psychiatric disease
* Severe or clinically significant cardiovascular disease uncontrolled with standard treatment
* Active systemic infections (including TB, pneumonia, Pneumocystis pneumonia, sepsis, and opportunistic infections)
* Parasitic infection: Subjects with a known parasitic infestation within 6 months prior to screening.
* HIV positive status
* Active hepatitis due to hepatitis B virus or hepatitis C virus
* Known history or presence of venous thromboembolism/venous thrombotic events (deep vein thrombosis and/or pulmonary embolus)
* laboratory parameter exclusions:

  1. Estimated glomerular filtration rate of <30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equations
  2. WBC count <4 × 109/L
  3. Absolute lymphocyte count <500 cells/mm3
  4. Absolute neutrophil count <1000 cells/mm3
  5. Platelet count <120,000/mm3
  6. Hemoglobin <8 g/dL (<80 g/L)
* Subjects who are pregnant, breastfeeding, or planning to become pregnant during the time of study participation
* History of clinically significant drug or alcohol abuse within the last 6 months
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in remission [OGC 4.0] | From Baseline to week 28
  The proportion of subjects in remission (oral glucocorticoid [OGC] 4.0) at Week 28 of the study treatment period.
  Definition of remission (OGC 4.0): BVAS of 0 AND OGC dose of prednisolone/prednisone ≤4 mg/day

SECONDARY OUTCOMES:
The proportion of subjects in remission [OGC 7.5] | From Baseline to week 28
  The proportion of subjects in remission (OGC 7.5) at Week 28 of the study treatment period Definition of remission (OGC 7.5): BVAS of 0 AND OGC dose of prednisolone/prednisone ≤7.5 mg/day
Time to first relapse of EGPA | Up to Week 28
  Relapse of EGPA will be defined as active disease since the last visit after remission (OGC 4.0) was achieved, characterized by:
  1. Active vasculitis (BVAS of >0); OR
  2. Signs and/or symptoms of active asthma with a corresponding worsening in answers on the 6-item Asthma Control Questionnaire (compared with the most recent previous results); OR
  3. Active nasal and/or sinus disease (attributable to EGPA) with a corresponding worsening in at least 1 of the answers on the sinonasal symptom questionnaire (compared with the most recent previous assessment).
Time to first worsening of EGPA | Up to Week 28
  Worsening of EGPA will be defined as worsening of active disease since the last visit, characterized by:
  1. Active vasculitis (BVAS >0) and the score greater than the previous visit; OR
  2. Signs and/or symptoms of active asthma with a corresponding worsening in answers on the 6-item Asthma Control Questionnaire (compared to the most recent previous score); OR
  3. Active nasal and/or sinus disease (attributable to EGPA) with a corresponding worsening in at least 1 of the answers on the sinonasal symptom questionnaire (compared to the most recent previous assessment).

CONTACTS AND LOCATIONS:
Locations (34):
- United States (7):
  - National Jewish Health, Denver, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - University of Toronto, Toronto, Ontario
- France (3):
  - CHU Nice, Nice
  - Hopital Cochin, Paris
  - Chu Rangueil, Toulouse
- Medius Kliniken gGmbh, Kirchheim unter Teck, Studienzentrale, Germany
- Italy (4):
  - Istituto Auxologico Italiano IRCCS, Milan
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Azienda Provinciale per i Servizi Sanitari Provincia Autonoma Trento, Trento
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (11):
  - Chiba University Hospital, Chuo-ku, Chiba-shi, Chiba
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - NHO Sagamihara National Hospital, Sagamihara, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
- Spain (2):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Complejo Hospitalario de Navarra, Pamplona
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Edgbaston, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Royal Berkshire NHS Foundation Trust, Reading

IPD SHARING:
Plan to Share IPD: No
Submission to the FDA